CLINICAL TRIAL: NCT03690466
Title: Ultrasound Treatment of Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Device Feasibility
Other Study IDs: RHEUM-2018-26732
Record Dates: First submitted 2018-09-20; First posted 2018-10-01 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This will be a controlled, randomized, double-blinded trial of short-term (14 days) treatment with ultrasound stimulation (therapeutic energy dose) or sham (no energy dose) delivered to the spleen.
  Participants will be provided a portable ultrasound device or sham device for at home use. Participants will be trained on how to use the device and will be instructed to use it for 30 minutes per day, at approximately the same time each day for 14 days.
  Participants will be assessed at several time points before, during and at the end of treatment as well as a one-week follow-up visit.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Study device treatment (Experimental): Transcutaneous non-invasive ultrasound will be administered to the spleen for 30 minutes every day for 2 weeks (14 days total) via a portable device.
  Interventions: Device: Study device treatment
- Sham device treatment (Sham Comparator): Sham treatment will be administered to the spleen for 30 minutes every day for 2 weeks (14 days total) via a portable device.
  Interventions: Device: Sham device treatment

INTERVENTIONS:
Device: Study device treatment — The ultrasound portable device comprises a tabletop control unit and a transducer connected to the control unit by a cord.
  Other Names: Treatment group
  Arms: Study device treatment
Device: Sham device treatment — A similar device as used for the study device treatment will be used, except that no energy will be delivered to the spleen.
  Other Names: Control group
  Arms: Sham device treatment

SUMMARY:
The research objective of the pilot study is to assess early feasibility of safety and efficacy of spleen ultrasound stimulation in the treatment of rheumatoid arthritis (RA) in a blinded and randomized controlled trial. Specific Aims include:

* Measure RA disease activity and functional/biomarker metrics during and after a 2- week course of spleen-directed daily ultrasound treatments (within-arm and between-arm assessments); and
* Monitor adverse events during and after daily ultrasound treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females aged 18 and over.
2. Must carry a diagnosis of rheumatoid arthritis, as defined by the American College of Rheumatology in 2010: (https://www.rheumatology.org/Portals/0/Files/2010_revised_criteria_classification_ra.pdf).

   Classification as "definite RA" is based on the confirmed presence of synovitis in at least one joint, absence of an alternative diagnosis that better explains the synovitis, and achievement of a total score of 6 or greater (of a possible 10) from the individual scores in 4 domains: number and site of involved joints (score range 0-5), serologic abnormality (score range 0-3), elevated acute-phase response (score range 0-1), and symptom duration (2 levels; range 0-1).
3. Exhibiting symptoms or signs of inadequate disease control according to one of 2 measures:

   Modified HAQ score of greater than 0.3 and DAS28-CRP greater than 3.2 (http://www.phusewiki.org/wiki/index.php?title=Disease_Activity_Score_-_CRP_(DAS-CRP).
4. Participants should have home access to broadband internet, such that online video conversations can occur with study personnel via study-provided personal digital assistive devices.

Exclusion Criteria:

1. Active bacterial or viral infection.
2. Pregnant women or presence of active malignancy.
3. Inability to perform minimal daily self-cares associated with feeding/dressing, according to HAQ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Within-arm change in the Disease Activity Score (DAS-28) from baseline to end of treatment for treatment group. | Day 0 (baseline) to Day 14 (end of treatment)
  Full p-value of 0.05 will be allocated to Primary Outcome Measure and then if outcome is satisfied, the full p-value of 0.05 will be allocated to Secondary Outcome Measure.

SECONDARY OUTCOMES:
Between-arm change in the DAS-28 from baseline to end of treatment. | Day 0 (baseline) to Day 14 (end of treatment)
  Full p-value of 0.05 will be allocated to Primary Outcome Measure and then if outcome is satisfied, the full p-value of 0.05 will be allocated to Secondary Outcome Measure.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Peterson, MD PHD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Goggins E, Inoue H, Okusa MD. Neuroimmune Control of Inflammation in Acute Kidney Injury and Multiorgan Dysfunction. J Am Soc Nephrol. 2025 Dec 1;36(12):2473-2484. doi: 10.1681/ASN.0000000813. Epub 2025 Jul 7. PMID 40622772